CLINICAL TRIAL: NCT00471068
Title: Study of Travatan and Cosopt in Primary Open-Angle Glaucoma or Ocular Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Question raised by Ethics Committee
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMD-05-03
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Results first posted 2010-01-08 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2010-02

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; dorzolamide-timolol combination; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travatan (Experimental): Travatan: 6 weeks treatment with Travatan (travoprost 40 mg/ml eye drops, solution) once daily at 08:00 and placebo (timolol vehicle) once daily at 20:00 in the affected eye(s)
  Interventions: Drug: Travatan; Drug: Placebo (Timolol Vehicle)
- Cosopt (Active Comparator): treatment period of 6 weeks with Cosopt (dorzolamide 20 mg/ml and timolol maleate 5 mg/ml eye drops, solution) twice daily at 08:00 and 20:00 in the affected eye(s)
  Interventions: Drug: Cosopt

INTERVENTIONS:
Drug: Travatan — Travatan: 6 weeks treatment with Travatan (travoprost 40 mg/ml eye drops, solution) once daily at 08:00 and placebo (timolol vehicle) once daily at 20:00 in the affected eye(s)
  Arms: Travatan
Drug: Cosopt — treatment period of 6 weeks with Cosopt (dorzolamide 20 mg/ml and timolol maleate 5 mg/ml eye drops, solution) twice daily at 08:00 and 20:00 in the affected eye(s)
  Arms: Cosopt
Drug: Placebo (Timolol Vehicle) — Travatan group: 6 weeks treatment with Travatan (travoprost 40 mg/ml eye drops, solution) once daily at 08:00 and placebo (timolol vehicle) once daily at 20:00 in the affected eye(s)
  Arms: Travatan

SUMMARY:
To compare the efficacy and safety in patients treated with travoprost versus dorzolamide/timolol maleate combination in patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patient with open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* By Age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grau, Study Director — Alcon Research
Locations (1):
- Coimbra, Coimbra, Portugal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: from 13-03-2007 to 30-11-2007 Recruitment restarted on 27-03-2008 to 27-05-2008 First patient first visit: 19-03-2007 Last patient last visit: 29-05-2008
Pre-assignment Details: After completing the run-in, 8 patients were not randomized: 7 patients did not meet entry criteria and 1 patient was excluded by sponsor's decision.
Period: Overall Study
Arm/Group | Travatan | Cosopt
Started | 21 | 25
Completed | 20 | 24
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travatan | Cosopt | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 16 | 26
  >=65 years | 11 | 9 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 7 | 15 | 22

OUTCOME MEASURES:

1. Primary Outcome: Intaocular Pressure (IOP) Mean Change After 6 Weeks of Treatment
Description: IOP measured at week 6 minus IOP measured at baseline
Time Frame: At week 0 and week 6
Measure: Mean (Standard Deviation); unit: millimeters mercury (mm Hg)
Arm/Group | Travatan | Cosopt
Number analyzed (Participants) | 21 | 25
millimeters mercury (mm Hg) | -4.57 (1.62) | -4.08 (2.50)

ADVERSE EVENTS:
Time Frame: Run-in (2-4 weeks) + treatment period (6 weeks)
Arm/Group | Travatan | Cosopt
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/25
Other Adverse Events (participants affected / at risk) | 2/21 | 3/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travatan (N=21) | Cosopt (N=25)
Inguinal hernia surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — This SAE occurred while patient was in the run-in period taking timolol
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travatan (N=21) | Cosopt (N=25)
Flu (Infections and infestations) | 0 (0) | 1 (1)
Ocular pruritus (Eye disorders) | 1 (1) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Redness eye (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Sample size smaller than the one defined by the protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No